CLINICAL TRIAL: NCT01226524
Title: The Role of Traditional Chinese Medicine in the Treatment of Chronic Childhood Immune Thrombocytopenia (ITP)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Shoshana Vilk, Prof. Shoshana Revel-Villk, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITP-HMO-CTIL
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2011-03

CONDITIONS: Childhood Chronic Immune Thrombocytopenia
MeSH Terms: interventions — bu-zhong-yi-qi-tang

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Traditional Chinese Medicine (Experimental): A traditional Chinese Medicine (TCM) therapist will diagnose and prescribe the herbal remedies according to TCM principles from one of four formulations or any combination of the four formulations, i.e. Bu Zhong Yi Qi Tang, Zhi Xue Tang, Chuan xin lian kang yan pian mod, Tian Wang Bu xin Dan
  Interventions: Drug: Bu Zhong Yi Qi Tang, Zhi Xue Tang, Chuan xin lian kang yan pian mod, Tian Wang Bu xin Dan

INTERVENTIONS:
Drug: Bu Zhong Yi Qi Tang, Zhi Xue Tang, Chuan xin lian kang yan pian mod, Tian Wang Bu xin Dan — A traditional Chinese Medicine (TCM) therapist will diagnose and prescribe the herbal remedies according to TCM principles from one of four formulations or any combination of the four formulation

SUMMARY:
Immune thrombocytopenia (ITP) is an autoimmune disorder manifested as isolated low platelet count which results in a tendency for bleeding. Around 10% of childhood ITP does not reach resolution within 1 year thus becoming chronic ITP. Therapeutic modalities at present are aimed to achieve symptomatic relief, do not change the natural course of the disorder and are associated with potential side effects and increase cost. Thus, identifying a new therapy that would decrease the bleeding symptoms, without causing significant adverse effects, could be very beneficial. Preliminary reports demonstrate a beneficial role for Traditional Chinese medicine (TCM) in the treatment of ITP.

Working hypothesis and aims: The use of TCM will improve the status of children with chronic ITP and thus will reduce the need to use conventional medications. The investigators aim to study whether in children with chronic ITP, supplementation with TCM, improves the bleeding symptoms and ITP-related quality of life (QOL) compared to the period prior to the intervention? Methods: The study includes three periods: 1st observation period (1 month), TMC period (3 months) and 2nd observation period (2 months). During all study periods the following data will be collected: bleeding symptoms, bleeding score, platelet count, need for conventional therapy, side effects of therapy and ITP-related QOL.

ELIGIBILITY:
Inclusion Criteria:

1. Children (< 18 years) diagnosed with chronic ITP; >1 year after a first diagnosis and baseline platelet count < 30,000. The diagnosis of ITP will be the responsibility of the Pediatric Hematology specialist in each participating center.

-

Exclusion Criteria:

1. Children with thrombocytopenia due to other causes. 2. Refusal of child or guardian to participate.

-

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2011-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To determine whether in children with chronic ITP, does supplementation with Traditional Chinese Medicine remedies, reduces symptomatic bleeding episodes compared to the period prior to intervention? | three month

SECONDARY OUTCOMES:
To determine whether in children with chronic ITP, does supplementation with TCM remedies, improves the disease related quality of life compared to the period prior to intervention? | three months

CONTACTS AND LOCATIONS:
Overall Officials: Shoshana Revel-Vilk, MD, MSc, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel